CLINICAL TRIAL: NCT05705700
Title: Biomarker Study Targeting Abiraterone Metabolites and Polymporphisms in Men With PSA Progression on Abiraterone for the Treatment of Castration Resistant or Castration Sensitive Prostate Cancer (The Bio-STAMP Study)
Brief Title: Biomarker Study of in Men With PSA Progression on Abi for CR or CS PC (Bio-STAMP)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Feasibility
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019LS229
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride; abiraterone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1245c positive (1245c+) patients with dutasteride (Experimental): Continue on abiraterone 1000 mg PO daily with dutasteride 3.5 mg PO daily as an add-on therapy until radiographic progression is documented
  Interventions: Drug: Dutasteride; Drug: Abiraterone
- 1245c positive (1245c+) patients (Experimental): Continue on abiraterone 1000 mg PO daily (the standard of care for PSA only progression) until radiographic progression is documented
  Interventions: Drug: Abiraterone
- 1245c negative (1245c-) patients (Experimental): abiraterone 1000 mg PO daily (the standard of care for PSA only progression) until radiographic progression is documented
  Interventions: Drug: Abiraterone

INTERVENTIONS:
Drug: Dutasteride — High dose Dutasteride (3.5 mg daily) as add-on therapy at time of PSA progression
  Other Names: Abiraterone
  Arms: 1245c positive (1245c+) patients with dutasteride
Drug: Abiraterone — 1000 mg PO daily
  Other Names: Dutasteride

SUMMARY:
This is a multicenter, Phase II randomized biomarker-based therapeutic study in metastatic prostate cancer experiencing prostate specific antigen (PSA) only progression (without visceral, bone or lymph node progression) while on abiraterone therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological evidence of adenocarcinoma of the prostate
* Undergone orchiectomy, or have been on luteinizing hormone-releasing hormone (LHRH) agonists or antagonists for at least 3 months prior to study enrollment. Patients on LHRH agonists/antagonists must remain on these agents for the duration of the study.
* Currently receiving abiraterone (ZYTIGA or FDA approved generic) in the castration sensitive (CSPC) or castration resistant (CRPC) setting with PSA progression in the absence of visceral, bone or lymph node progression. PSA progression is defined as an increase in the PSA level of more than 50% above the nadir with two consecutive increases at least 2 weeks apart (based on Prostate Cancer Working Group Criteria, version 3 (PCWG3).
* Minimum PSA must be ≥1.0 ng/dL.
* Age 18 years of age or older.
* ECOG performance status 0 or 1.
* Have adequate organ function confirmed by the following laboratory values obtained within 14 days prior to enrollment:

  * absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
  * platelets ≥ 100 × 10^9/L
  * hemoglobin ≥ 10 g/dL, independent of transfusion ≤14 days of screening
  * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN); if liver metastases, then ≤ 5 × ULN
  * total bilirubin ≤ 1.5 × ULN; < 2 × ULN if hyperbilirubinemia is due to Gilbert's syndrome
  * serum albumin ≥ 30 g/L (3.0 g/dL)
  * Serum creatinine ≤ 1.5 x ULN; OR estimated glomerular filtration rate (GFR) ≥ 45 mL/min using the Cockcroft Gault formula
* Participants with partners of childbearing potential must be willing to use at least two forms of effective birth control (one form must be a barrier method) during the dutasteride treatment period and for 6 months after last dose or 3 weeks after the last dose of abiraterone whichever is longer. Persons are considered to be of childbearing potential unless one or the following applies:

  * Is postmenopausal, defined as no menses for at least 12 months without an alternative medical cause
  * Considered permanently sterile. Permanent sterilization includes hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy.
* Voluntary written consent prior to the performance of any research related activit

Exclusion Criteria:

* Previously demonstrated, clinically significant hypersensitivity (e.g., serious skin reactions, angioedema) to 5 alpha-reductase inhibitors (i.e. finasteride).
* Prior use of Enzalutamide, Apalutamide, or Darolutamide for the treatment of prostate cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with radiographic progression free survival (rPFS) rate | 24 Weeks after study treatment
  Count the the number of patients with radiographic progression free survival (rPFS)

SECONDARY OUTCOMES:
Determine overall survival (OS) | 24 months from start of treatment assignment
  The Kaplan-Meier product-limit estimator will be used to estimate OS distribution
Number of patients with a PSA decline of ≥ 50% | 24 weeks of adding of adding high-dose dutasteride
  Count the number of patients with serologic progression. It is defined as an increase in the PSA level of more than 50% above the nadir with two consecutive increases confirmed at least 2 weeks apart.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ryan, MD, Principal Investigator — Masonic Cancer Center, Univeristy of Minnesota

IPD SHARING:
Plan to Share IPD: No